CLINICAL TRIAL: NCT01136421
Title: Magnesium Sulfate Versus Ipratropuim Bromide in Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: State secretary of research, High education and research ministery
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Magnesium sulfate
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-05

CONDITIONS: COPD Exacerbation
Keywords: COPD exacerbation; Magnesium sulfate; Ipratropium bromide; Emergency departement
MeSH Terms: interventions — Ipratropium; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ipratropium bromide (Active Comparator): Patients received ipratropium bromide (IB group, 0.5 mg in 3 mL of normal saline) delivered via aerosol mask at 10 L/min driven by pressurised air. Simultaneously, patients received intravenous placebo (10 mL of normal saline). Thereafter 4 doses of nebulised IB with terbutaline are administered at 30 min intervals.
  Interventions: Drug: Ipratropium bromide
- Magnesium sulfate (Experimental): Patients received magnesium sulfate (MgSO4 group, 150 mg in 4 mL of normal saline)delivered via aerosol mask at 10 L/min driven by pressurised air. Simultaneously, additional magnesium sulfate is given as an intravenous bolus (1.5g in 10 ml). Patients received thereafter 4 doses of nebulized magnesium sulfate with terbutaline at 30 min intervals.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Ipratropium bromide — Patients received ipratropium bromide (IB group, 0.5 mg in 3 mL of normal saline) delivered via aerosol mask at 10 L/min driven by pressurised air. Simultaneously, patients received intravenous placebo (10 mL of normal saline). Thereafter 4 doses of nebulised IB with terbutaline are administered at 30 min intervals.
  Arms: Ipratropium bromide
Drug: Magnesium Sulfate — Patients received magnesium sulfate (MgSO4 group, 150 mg in 4 mL of normal saline)delivered via aerosol mask at 10 L/min driven by pressurised air. Simultaneously, additional magnesium sulfate is given as an intravenous bolus (1.5g in 10 ml). Patients received thereafter 4 doses of nebulized magnesium sulfate with terbutaline at 30 min intervals.
  Arms: Magnesium sulfate

SUMMARY:
Treatment with short acting β2 agonists for exacerbations of COPD results in clinical improvement. It has not been established whether combining short acting β2 agonists to other bronchodilators is more effective than β2 agonists alone. The aim of this study is to evaluate the efficacy and safety of combination of SABA and MgSO4 in comparison to SABA and ipratropium bromide (IB) in patients attending the emergency department for AECOPD.

DETAILED DESCRIPTION:
Patients presenting to the emergency department with exacerbation of COPD are randomized to receive nebulised ipratropuim bromide or combined nebulised and an intravenous bolus of magnesium sulfate during 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* 40 years old or over
* have known or suspected COPD based on pulmonary function test, arterial blood gas, clinical history, physical examination, and chest radiograph
* worsening of dyspnea within 2 weeks,
* partial pressure of arterial carbon dioxide (PaCO2) >45 mmHg
* respiratory rate >24/min
* arterial pH <7.35
* partial pressure of arterial oxygen (PaO2) <50 mmHg under room air

Exclusion Criteria:

* hypersensitivity to anticholinergics and to magnesium sulfate
* patients that received anticholinergics within 6 hours before ED admission
* systolic arterial pressure <90 mmHg or need to vasoactive drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: semir nouira, Pr, Principal Investigator — University of Monastir
Locations (2):
- Tunisia (2):
  - University Hospital of Monastir, Monastir, Monstir
  - Soudani Marghli, Mahdia, Tunisia